CLINICAL TRIAL: NCT04270136
Title: Feasibility of Total Mastectomy in Ambulatory Care
Acronym: AMASTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Beauvais (Other); Centre Hospitalier de Saint-Quentin (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0061
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Mastectomy; Ambulatory Care
Keywords: Breast Cancer; mastectomy; ambulatory care
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Simple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- breast cancer mastectomy (Experimental)
  Interventions: Procedure: total mastectomy

INTERVENTIONS:
Procedure: total mastectomy — breast cancer non conserving surgery

SUMMARY:
Breast cancer is the first female cancer in France. Total mastectomy occurred in 30% of breast cancer patient population.

The purpose of this study is to evaluate the feasibility of outpatient surgery for the total mastectomy.

In France, Ambulatory care is developed as part of the new national health plan.

Breast conserving surgery for tumorectomy or partial mastectomy is already done in outpatient vacation.

Total mastectomy is an extension of this surgery, and, as such, underpins the investigator's hypothesis that total mastectomy is feasible in outpatient care .

ELIGIBILITY:
Inclusion Criteria:

* All patient with an indication of breast non conserving surgery

Exclusion Criteria:

* Standard contra-indication for ambulatory care.
* Also bilateral surgery and immediate breast reconstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female with breast cancer
Enrollment: 1 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
number of ambulatory care after total mastectomy allowed with PADSS score | day 0= day of surgery
  Post Anaesthetic Discharge Scoring System (PADSS), which considers six criteria: vital signs, ambulation, nausea/vomiting, pain, bleeding and voiding. Each criterion is given a score ranging from 0 to 2. Only patients who achieve a score of 9 or more are considered ready for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Demblocque, MD, Principal Investigator — Centre Hospitalier de Beauvais; Albine Mancaux, MD, Principal Investigator — Centre Hospitalier de Beauvais; Pierrick Theret, MD, Principal Investigator — CH SAINT-QUENTIN
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No